CLINICAL TRIAL: NCT01945268
Title: A Randomized Controlled Trial of Influenza Vaccine to Prevent Adverse Vascular Events: A Pilot Study
Brief Title: Influenza Vaccine To Prevent Adverse Vascular Events:Pilot
Acronym: IVVE:Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCT IVVE Pilot
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: vascular, influenza, vaccine, heart failure
MeSH Terms: conditions — Heart Failure; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- influenza vaccine (Experimental): Participants at high risk for adverse vascular events will be immunized with 0.5 ml dose of inactivated trivalent influenza vaccine
  Interventions: Drug: inactivated trivalent influenza vaccine
- placebo vaccination (Placebo Comparator): Participants at high risk for adverse vascular events will be immunized with a 0.5 ml dose of sterile saline inactivated during the influenza season.
  Interventions: Other: Sterile saline

INTERVENTIONS:
Drug: inactivated trivalent influenza vaccine — 0.5 ml dose injected intramuscularly
  Other Names: VAXIGRIP vaccine
  Arms: influenza vaccine
Other: Sterile saline — 0.5 ml dose injected intramuscularly
  Arms: placebo vaccination

SUMMARY:
A multi-centre, randomized, placebo controlled, trial. Participants at high-risk for vascular events from the network of INTER- CHF will be randomized to inactivated influenza vaccine or placebo and followed prospectively over three influenza seasons. 600 participants will be enrolled prior to influenza season and randomized to either influenza vaccine or saline placebo.

DETAILED DESCRIPTION:
Cardiovascular disease is a major cause of morbidity and mortality. There is recent evidence that infection due to influenza may precipitate vascular events such as myocardial infarctions and strokes. There is some evidence that influenza vaccination may prevent such events but the data are inconclusive. The investigators propose a randomized controlled trial to assess whether influenza vaccination will prevent vascular illness. Adults with clinical heart failure will be randomized to inactivated influenza vaccine or saline placebo. This pilot study will provide needed data to establish the feasibility of a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and NYHA functional class II, III and IV

Exclusion Criteria:

* Anaphylactic reaction to a previous dose of TIV
* Known IgE-mediated hypersensitivity to eggs manifested as hives, swelling of the mouth and throat, difficulty in breathing, hypotension, or shock
* Guillain-Barré syndrome within eight weeks of a previous influenza vaccine
* Anaphylactic reaction to neomycin
* Patients who have had influenza vaccine in two of the three previous years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | Six months
  If no more than 5% of all recruited subjects crossed over from one study group to the other, and if there is at least 98% follow up.

SECONDARY OUTCOMES:
Adverse cardiovascular event | Six months
  The primary outcome will be a composite of cardiovascular death, non-fatal myocardial infarction, non-fatal stroke and hospitalizations for heart failure using standardized criteria.
Cardiovascular death | Six months
  CV death alone will be a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, MSc, Principal Investigator — McMaster University
Locations (3):
- Maputo Central Hospital, Maputo, Mozambique
- University of Philippines, Manila, Emita, Philippines
- Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DataFax - Data Management Software for Clinical Trials. http://www.datafax.com/; accessed February 15, 2013.
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] ACCORD Study Group; Cushman WC, Evans GW, Byington RP, Goff DC Jr, Grimm RH Jr, Cutler JA, Simons-Morton DG, Basile JN, Corson MA, Probstfield JL, Katz L, Peterson KA, Friedewald WT, Buse JB, Bigger JT, Gerstein HC, Ismail-Beigi F. Effects of intensive blood-pressure control in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1575-85. doi: 10.1056/NEJMoa1001286. Epub 2010 Mar 14. PMID 20228401
- [Background] ACCORD Study Group; Ginsberg HN, Elam MB, Lovato LC, Crouse JR 3rd, Leiter LA, Linz P, Friedewald WT, Buse JB, Gerstein HC, Probstfield J, Grimm RH, Ismail-Beigi F, Bigger JT, Goff DC Jr, Cushman WC, Simons-Morton DG, Byington RP. Effects of combination lipid therapy in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1563-74. doi: 10.1056/NEJMoa1001282. Epub 2010 Mar 14. PMID 20228404
- [Background] CURRENT-OASIS 7 Investigators; Mehta SR, Bassand JP, Chrolavicius S, Diaz R, Eikelboom JW, Fox KA, Granger CB, Jolly S, Joyner CD, Rupprecht HJ, Widimsky P, Afzal R, Pogue J, Yusuf S. Dose comparisons of clopidogrel and aspirin in acute coronary syndromes. N Engl J Med. 2010 Sep 2;363(10):930-42. doi: 10.1056/NEJMoa0909475. PMID 20818903
- [Background] ACCORD Study Group; Gerstein HC, Miller ME, Genuth S, Ismail-Beigi F, Buse JB, Goff DC Jr, Probstfield JL, Cushman WC, Ginsberg HN, Bigger JT, Grimm RH Jr, Byington RP, Rosenberg YD, Friedewald WT. Long-term effects of intensive glucose lowering on cardiovascular outcomes. N Engl J Med. 2011 Mar 3;364(9):818-28. doi: 10.1056/NEJMoa1006524. PMID 21366473
- [Background] ORIGIN Trial Investigators; Bosch J, Gerstein HC, Dagenais GR, Diaz R, Dyal L, Jung H, Maggiono AP, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. n-3 fatty acids and cardiovascular outcomes in patients with dysglycemia. N Engl J Med. 2012 Jul 26;367(4):309-18. doi: 10.1056/NEJMoa1203859. Epub 2012 Jun 11. PMID 22686415
- [Background] ORIGIN Trial Investigators; Gerstein HC, Bosch J, Dagenais GR, Diaz R, Jung H, Maggioni AP, Pogue J, Probstfield J, Ramachandran A, Riddle MC, Ryden LE, Yusuf S. Basal insulin and cardiovascular and other outcomes in dysglycemia. N Engl J Med. 2012 Jul 26;367(4):319-28. doi: 10.1056/NEJMoa1203858. Epub 2012 Jun 11. PMID 22686416
- [Background] Ontario Case Costing Initiative. Toronto, Ontario: Ontario Ministry of Health and Long-term Care, 2005. (Accessed January 29, 2011 at http://www.occp.com).
- [Background] Brown PD, Lerner SA. Community-acquired pneumonia. Lancet. 1998 Oct 17;352(9136):1295-302. doi: 10.1016/S0140-6736(98)02239-9. PMID 9788476
- [Background] Call SA, Vollenweider MA, Hornung CA, Simel DL, McKinney WP. Does this patient have influenza? JAMA. 2005 Feb 23;293(8):987-97. doi: 10.1001/jama.293.8.987. PMID 15728170
- [Background] Einhorn PT, Davis BR, Massie BM, Cushman WC, Piller LB, Simpson LM, Levy D, Nwachuku CE, Black HR; ALLHAT Collaborative Research Group. The Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) Heart Failure Validation Study: diagnosis and prognosis. Am Heart J. 2007 Jan;153(1):42-53. doi: 10.1016/j.ahj.2006.10.012. PMID 17174636
- [Background] Granger CB, Vogel V, Cummings SR, Held P, Fiedorek F, Lawrence M, Neal B, Reidies H, Santarelli L, Schroyer R, Stockbridge NL, Feng Zhao. Do we need to adjudicate major clinical events? Clin Trials. 2008;5(1):56-60. doi: 10.1177/1740774507087972. PMID 18283081
- [Background] Pogue J, Walter SD, Yusuf S. Evaluating the benefit of event adjudication of cardiovascular outcomes in large simple RCTs. Clin Trials. 2009 Jun;6(3):239-51. doi: 10.1177/1740774509105223. PMID 19528133
- [Background] Djulbegovic B, Lacevic M, Cantor A, Fields KK, Bennett CL, Adams JR, Kuderer NM, Lyman GH. The uncertainty principle and industry-sponsored research. Lancet. 2000 Aug 19;356(9230):635-8. doi: 10.1016/S0140-6736(00)02605-2. PMID 10968436
- [Background] Canadian Community Health Survey: influenza immunization coverage results. http://www.bccdc.ca/imm-vac/BCImmunizationCov/flucoverage/default.htm.
- [Background] Mereckiene J, Cotter S, Nicoll A, Levy-Bruhl D, Ferro A, Tridente G, Zanoni G, Berra P, Salmaso S, O'Flanagan D, O Flanagan D; VENICE Project Gatekeepers Group. National seasonal influenza vaccination survey in Europe, 2008. Euro Surveill. 2008 Oct 23;13(43):19017. doi: 10.2807/ese.13.43.19017-en. PMID 18947524
- [Background] Blank PR, Schwenkglenks M, Szucs TD. Disparities in influenza vaccination coverage rates by target group in five European countries: trends over seven consecutive seasons. Infection. 2009 Oct;37(5):390-400. doi: 10.1007/s15010-009-8467-y. Epub 2009 Sep 18. PMID 19768382
- [Background] Centers for Disease Control and Prevention (CDC). Prevention and control of influenza with vaccines: recommendations of the Advisory Committee on Immunization Practices (ACIP)--United States, 2012-13 influenza season. MMWR Morb Mortal Wkly Rep. 2012 Aug 17;61(32):613-8. PMID 22895385
- [Background] Canadian Communicable Disease Report 2012. Statement on seasonal influenza vaccine for 2012-2013; 38: 2012.
- [Background] Natarajan P, Cannon CP. Myocardial infarction vaccine? Evidence supporting the influenza vaccine for secondary prevention. Eur Heart J. 2011 Jul;32(14):1701-3. doi: 10.1093/eurheartj/ehr053. Epub 2011 Mar 15. No abstract available. PMID 21406438
- [Background] Phrommintikul A, Kuanprasert S, Wongcharoen W, Kanjanavanit R, Chaiwarith R, Sukonthasarn A. Influenza vaccination reduces cardiovascular events in patients with acute coronary syndrome. Eur Heart J. 2011 Jul;32(14):1730-5. doi: 10.1093/eurheartj/ehr004. Epub 2011 Feb 2. PMID 21289042
- [Background] Ciszewski A, Bilinska ZT, Brydak LB, Kepka C, Kruk M, Romanowska M, Ksiezycka E, Przyluski J, Piotrowski W, Maczynska R, Ruzyllo W. Influenza vaccination in secondary prevention from coronary ischaemic events in coronary artery disease: FLUCAD study. Eur Heart J. 2008 Jun;29(11):1350-8. doi: 10.1093/eurheartj/ehm581. Epub 2008 Jan 10. PMID 18187561
- [Background] Gurfinkel EP, Leon de la Fuente R, Mendiz O, Mautner B. Flu vaccination in acute coronary syndromes and planned percutaneous coronary interventions (FLUVACS) Study. Eur Heart J. 2004 Jan;25(1):25-31. doi: 10.1016/j.ehj.2003.10.018. PMID 14683739
- [Background] Warren-Gash C, Smeeth L, Hayward AC. Influenza as a trigger for acute myocardial infarction or death from cardiovascular disease: a systematic review. Lancet Infect Dis. 2009 Oct;9(10):601-10. doi: 10.1016/S1473-3099(09)70233-6. PMID 19778762
- [Background] Keller T, Weeda VB, van Dongen CJ, Levi M. Influenza vaccines for preventing coronary heart disease. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD005050. doi: 10.1002/14651858.CD005050.pub2. PMID 18646119
- [Background] Population Health Research Institute http://www.phri.ca/
- [Background] Jackson LA, Nelson JC, Benson P, Neuzil KM, Reid RJ, Psaty BM, Heckbert SR, Larson EB, Weiss NS. Functional status is a confounder of the association of influenza vaccine and risk of all cause mortality in seniors. Int J Epidemiol. 2006 Apr;35(2):345-52. doi: 10.1093/ije/dyi275. Epub 2005 Dec 20. PMID 16368724
- [Background] Jackson LA, Jackson ML, Nelson JC, Neuzil KM, Weiss NS. Evidence of bias in estimates of influenza vaccine effectiveness in seniors. Int J Epidemiol. 2006 Apr;35(2):337-44. doi: 10.1093/ije/dyi274. Epub 2005 Dec 20. PMID 16368725
- [Background] Telmisartan Randomised AssessmeNt Study in ACE iNtolerant subjects with cardiovascular Disease (TRANSCEND) Investigators; Yusuf S, Teo K, Anderson C, Pogue J, Dyal L, Copland I, Schumacher H, Dagenais G, Sleight P. Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial. Lancet. 2008 Sep 27;372(9644):1174-83. doi: 10.1016/S0140-6736(08)61242-8. Epub 2008 Aug 29. PMID 18757085
- [Background] ONTARGET Investigators; Yusuf S, Teo KK, Pogue J, Dyal L, Copland I, Schumacher H, Dagenais G, Sleight P, Anderson C. Telmisartan, ramipril, or both in patients at high risk for vascular events. N Engl J Med. 2008 Apr 10;358(15):1547-59. doi: 10.1056/NEJMoa0801317. Epub 2008 Mar 31. PMID 18378520
- [Background] Teo K, Yusuf S, Sleight P, Anderson C, Mookadam F, Ramos B, Hilbrich L, Pogue J, Schumacher H; ONTARGET/TRANSCEND Investigators. Rationale, design, and baseline characteristics of 2 large, simple, randomized trials evaluating telmisartan, ramipril, and their combination in high-risk patients: the Ongoing Telmisartan Alone and in Combination with Ramipril Global Endpoint Trial/Telmisartan Randomized Assessment Study in ACE Intolerant Subjects with Cardiovascular Disease (ONTARGET/TRANSCEND) trials. Am Heart J. 2004 Jul;148(1):52-61. doi: 10.1016/j.ahj.2004.03.020. PMID 15215792
- [Background] Johnstone J, Loeb M, Teo KK, Gao P, Dyal L, Liu L, Avezum A, Cardona-Munoz E, Sleight P, Fagard R, Yusuf S; Ongoing Telmisartan Alone and in Combination With Ramipril Global EndPoint Trial (ONTARGET); Telmisartan Randomized Assessment Study in ACE Intolerant Subjects With Cardiovascular Disease (TRANSCEND) Investigators. Influenza vaccination and major adverse vascular events in high-risk patients. Circulation. 2012 Jul 17;126(3):278-86. doi: 10.1161/CIRCULATIONAHA.111.071100. Epub 2012 Jun 19. PMID 22715472
- [Background] Wang CS, Wang ST, Lai CT, Lin LJ, Chou P. Impact of influenza vaccination on major cause-specific mortality. Vaccine. 2007 Jan 26;25(7):1196-203. doi: 10.1016/j.vaccine.2006.10.015. Epub 2006 Oct 25. PMID 17097773
- [Background] Armstrong BG, Mangtani P, Fletcher A, Kovats S, McMichael A, Pattenden S, Wilkinson P. Effect of influenza vaccination on excess deaths occurring during periods of high circulation of influenza: cohort study in elderly people. BMJ. 2004 Sep 18;329(7467):660. doi: 10.1136/bmj.38198.594109.AE. Epub 2004 Aug 15. PMID 15313884
- [Background] Jackson LA, Yu O, Heckbert SR, Psaty BM, Malais D, Barlow WE, Thompson WW; Vaccine Safety Datalink Study Group. Influenza vaccination is not associated with a reduction in the risk of recurrent coronary events. Am J Epidemiol. 2002 Oct 1;156(7):634-40. doi: 10.1093/aje/kwf073. PMID 12244032
- [Background] Nichol KL, Nordin J, Mullooly J, Lask R, Fillbrandt K, Iwane M. Influenza vaccination and reduction in hospitalizations for cardiac disease and stroke among the elderly. N Engl J Med. 2003 Apr 3;348(14):1322-32. doi: 10.1056/NEJMoa025028. PMID 12672859
- [Background] Heffelfinger JD, Heckbert SR, Psaty BM, Weiss NS, Thompson WW, Bridges CB, Jackson LA. Influenza vaccination and risk of incident myocardial infarction. Hum Vaccin. 2006 Jul-Aug;2(4):161-6. doi: 10.4161/hv.2.4.2943. Epub 2006 Jul 24. PMID 17012887
- [Background] Siriwardena AN, Gwini SM, Coupland CA. Influenza vaccination, pneumococcal vaccination and risk of acute myocardial infarction: matched case-control study. CMAJ. 2010 Oct 19;182(15):1617-23. doi: 10.1503/cmaj.091891. Epub 2010 Sep 20. PMID 20855479
- [Background] Siscovick DS, Raghunathan TE, Lin D, Weinmann S, Arbogast P, Lemaitre RN, Psaty BM, Alexander R, Cobb LA. Influenza vaccination and the risk of primary cardiac arrest. Am J Epidemiol. 2000 Oct 1;152(7):674-7. doi: 10.1093/aje/152.7.674. PMID 11032163
- [Background] Lavallee P, Perchaud V, Gautier-Bertrand M, Grabli D, Amarenco P. Association between influenza vaccination and reduced risk of brain infarction. Stroke. 2002 Feb;33(2):513-8. doi: 10.1161/hs0202.102328. PMID 11823662
- [Background] Meyers D, Beahm D, Jurisich P, Milford C, Edlavich S. Influenza and pneumococcal vaccinations fail to prevent myocardial infarction. Heart Drug. 2004;4:96 -100.
- [Background] Remme WJ, Torp-Pedersen C, Cleland JG, Poole-Wilson PA, Metra M, Komajda M, Swedberg K, Di Lenarda A, Spark P, Scherhag A, Moullet C, Lukas MA. Carvedilol protects better against vascular events than metoprolol in heart failure: results from COMET. J Am Coll Cardiol. 2007 Mar 6;49(9):963-71. doi: 10.1016/j.jacc.2006.10.059. Epub 2007 Feb 20. PMID 17336720
- [Background] Naghavi M, Barlas Z, Siadaty S, Naguib S, Madjid M, Casscells W. Association of influenza vaccination and reduced risk of recurrent myocardial infarction. Circulation. 2000 Dec 19;102(25):3039-45. doi: 10.1161/01.cir.102.25.3039. PMID 11120692
- [Background] Gwini SM, Coupland CA, Siriwardena AN. The effect of influenza vaccination on risk of acute myocardial infarction: self-controlled case-series study. Vaccine. 2011 Feb 1;29(6):1145-9. doi: 10.1016/j.vaccine.2010.12.017. Epub 2010 Dec 18. PMID 21172383
- [Background] Kawano H, Motoyama T, Hirashima O, Hirai N, Miyao Y, Sakamoto T, Kugiyama K, Ogawa H, Yasue H. Hyperglycemia rapidly suppresses flow-mediated endothelium-dependent vasodilation of brachial artery. J Am Coll Cardiol. 1999 Jul;34(1):146-54. doi: 10.1016/s0735-1097(99)00168-0. PMID 10400004
- [Background] Lundman P, Eriksson M, Schenck-Gustafsson K, Karpe F, Tornvall P. Transient triglyceridemia decreases vascular reactivity in young, healthy men without risk factors for coronary heart disease. Circulation. 1997 Nov 18;96(10):3266-8. doi: 10.1161/01.cir.96.10.3266. PMID 9396413
- [Background] Conti CR. Vascular events responsible for thrombotic occlusion of a blood vessel. Clin Cardiol. 1993 Nov;16(11):761-2. doi: 10.1002/clc.4960161103. PMID 8269651
- [Background] Wanishsawad C, Zhou YF, Epstein SE. Chlamydia pneumoniae-induced transactivation of the major immediate early promoter of cytomegalovirus: potential synergy of infectious agents in the pathogenesis of atherosclerosis. J Infect Dis. 2000 Feb;181(2):787-90. doi: 10.1086/315235. PMID 10669378
- [Background] Davies MJ. The composition of coronary-artery plaques. N Engl J Med. 1997 May 1;336(18):1312-4. doi: 10.1056/NEJM199705013361809. No abstract available. PMID 9113937
- [Background] Chan NN, Colhoun HM, Vallance P. Cardiovascular risk factors as determinants of endothelium-dependent and endothelium-independent vascular reactivity in the general population. J Am Coll Cardiol. 2001 Dec;38(7):1814-20. doi: 10.1016/s0735-1097(01)01669-2. PMID 11738279
- [Background] Gheorghiade M, Bohm M, Greene SJ, Fonarow GC, Lewis EF, Zannad F, Solomon SD, Baschiera F, Botha J, Hua TA, Gimpelewicz CR, Jaumont X, Lesogor A, Maggioni AP; ASTRONAUT Investigators and Coordinators. Effect of aliskiren on postdischarge mortality and heart failure readmissions among patients hospitalized for heart failure: the ASTRONAUT randomized trial. JAMA. 2013 Mar 20;309(11):1125-35. doi: 10.1001/jama.2013.1954. PMID 23478743
- [Background] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Background] Swedberg K, Komajda M, Bohm M, Borer JS, Ford I, Dubost-Brama A, Lerebours G, Tavazzi L; SHIFT Investigators. Ivabradine and outcomes in chronic heart failure (SHIFT): a randomised placebo-controlled study. Lancet. 2010 Sep 11;376(9744):875-85. doi: 10.1016/S0140-6736(10)61198-1. PMID 20801500
- [Background] Homma S, Thompson JL, Pullicino PM, Levin B, Freudenberger RS, Teerlink JR, Ammon SE, Graham S, Sacco RL, Mann DL, Mohr JP, Massie BM, Labovitz AJ, Anker SD, Lok DJ, Ponikowski P, Estol CJ, Lip GY, Di Tullio MR, Sanford AR, Mejia V, Gabriel AP, del Valle ML, Buchsbaum R; WARCEF Investigators. Warfarin and aspirin in patients with heart failure and sinus rhythm. N Engl J Med. 2012 May 17;366(20):1859-69. doi: 10.1056/NEJMoa1202299. Epub 2012 May 2. PMID 22551105
- [Background] Warren-Gash C, Hayward AC, Hemingway H, Denaxas S, Thomas SL, Timmis AD, Whitaker H, Smeeth L. Influenza infection and risk of acute myocardial infarction in England and Wales: a CALIBER self-controlled case series study. J Infect Dis. 2012 Dec 1;206(11):1652-9. doi: 10.1093/infdis/jis597. Epub 2012 Oct 9. PMID 23048170
- [Background] Smeeth L, Thomas SL, Hall AJ, Hubbard R, Farrington P, Vallance P. Risk of myocardial infarction and stroke after acute infection or vaccination. N Engl J Med. 2004 Dec 16;351(25):2611-8. doi: 10.1056/NEJMoa041747. PMID 15602021
- [Background] Pesonen E, Andsberg E, Grubb A, Rautelin H, Meri S, Persson K, Puolakkainen M, Sarna S, Ohlin H. Elevated infection parameters and infection symptoms predict an acute coronary event. Ther Adv Cardiovasc Dis. 2008 Dec;2(6):419-24. doi: 10.1177/1753944708098695. PMID 19124438
- [Background] Guan XR, Li X, Xin XM, Jiang LX, Cui LY, Wang LF, Li HY. Influenza virus infection and risk of acute myocardial infarction. Inflammation. 2008 Aug;31(4):266-72. doi: 10.1007/s10753-008-9074-2. PMID 18568394
- [Background] Kinlay S, Ganz P. Role of endothelial dysfunction in coronary artery disease and implications for therapy. Am J Cardiol. 1997 Nov 6;80(9A):11I-16I. doi: 10.1016/s0002-9149(97)00793-5. PMID 9375937
- [Background] Zheng Z, Mittelman M, Tofler G, Pomeroy C, Dampier C, Wides B, Muller J. Infections prior to acute myocardial infarction onset. J Am Coll Cardiol. 1998;31(suppl 1):132-133.
- [Background] Tracking Heart Disease and Stroke in Canada. Released June 2009.
- [Background] Statistics Canada. Morality, Summary List of Causes 2008. Released October 18, 2011.
- [Background] Causes of death 2008, World Health Organization, Geneva, http://www.who.int/healthinfo/ global_burden_disease/ cod_2008_sources_methods.pdf.